CLINICAL TRIAL: NCT06091358
Title: Does a 4-week Inspiratory Muscle Training Intervention (IMT) Increase Inspiratory Muscle Pressure (MIP) and Other Functional Outcomes in People With Long COVID? A Pilot Investigation
Brief Title: Inspiratory Muscle Training in People With Long COVID-19- A Pilot Investigation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Rachel Eddy, Principle Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MSES 22/23-013-A1
Record Dates: First submitted 2023-10-18; First posted 2023-10-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Long COVID
Keywords: Dyspnea; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Dyspnea

STUDY DESIGN:
Intervention Model Description: Randomised parallel control group pilot investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will arrive at the Laboratory and complete a series of questionnaires: general physical activity, BDI, TDI, PSQI, General health questionnaire, Post COVID fatigue scale, EQ 5D-5L. They will undergo spirometry testing FEV1, MIP and PEF. Participants will undergo a 6 minute walk test and a Sub-maximal exercise test (CPET) using a cycle ergometer (15W/min) until an RPE of 17.
  Participants continue usual life between baseline and follow up testing. Participants will have 1 call per week where MIP is measured using a Care fusion hand held spirometer device.
  After 4 weeks, participants will return to the Laboratory and repeat baseline testing.
- Inspiratory Muscle training intervention (Experimental): Participants will arrive at the Laboratory and complete a series of questionnaires: general physical activity, BDI, TDI, PSQI, General health questionnaire, Post COVID fatigue scale, EQ 5D-5L. They will undergo spirometry testing FEV1, MIP and PEF. Participants will undergo a 6 minute walk test and a Sub-maximal exercise test (CPET) using a cycle ergometer (15W/min) until an RPE of 17.
  Participants undergo inspiratory muscle training for 4 weeks between baseline and follow up testing. They will be given a PrO2 device where the intervention will be 3 times per week for 4 weeks. Each session will be 6x6 breaths at 80% MIP. Participants will have 1 call per week where MIP is measured using a Care fusion hand held spirometer device.
  After 4 weeks, participants will return to the Laboratory and repeat baseline testing.
  Interventions: Device: PrO2

INTERVENTIONS:
Device: PrO2 — The intervention arm will receive a handheld PrO2 device and will participate in two unsupervised sessions and one supervised via Microsoft teams sessions per week.
  Participants will complete 3 sessions per week, for 4 weeks. Each session will include 6 x 6 inspirations at 80% of MIP. MIP will be measured on the supervised session day each week.
  Arms: Inspiratory Muscle training intervention

SUMMARY:
This pilot investigation will recruit people with Long COVID to participate in a 4 week individualized inspiratory muscle training intervention with pre and post spirometry testing and additional functional outcomes to assess the effectiveness of the intervention.

DETAILED DESCRIPTION:
The study design is a 4 - week parallel-arm intervention, randomised controlled trial. Participants will attend 2 testing days, baseline and follow-up 4 weeks apart.

Participants will first be screened over the phone to assess eligibility. Participants will then be randomly allocated using minimisation, into either control or intervention arm.

Baseline testing:

Participants will undergo baseline testing in the laboratory.

Participants will be measured for their anthropometrics; height and weight. Participants will complete a series of questionnaires for 15 mins.

Following 15 minutes rest, participants will then have three resting blood pressure and heart rate measurements and averaged via a sphygmomanometer and polar HR watch.

MIP will be measured using the MicroRPM care fusion 3 times and the highest value reported (10 minutes). Forced expiratory value in 1 second (FEV1) and peak expiratory flow (PEF) will be measured using Vitalograph 700 (Spirotrac 6).

Participants will undergo a 6-minute-walk-test self-paced where Rating of perceived exertion (RPE) and Borg dyspnea scale (BDS) will be assessed each minute. Then a sub-maximal exercise test using a cycle ergometer and VyntusCPX, where Ventilatory threshold (VT) and Maximal heart rate (HRMax)will be measured. Participants will be asked to cycle until they reach a 17 RPE on a ramp test of 10-15W/min (>20mins). Heart rate (HR), Rating percieved exertion (RPE) and Borg dyspnea scale BDS) measured each minute.

The intervention arm will receive a handheld PrO2 device and will participate in two unsupervised sessions and one supervised via Microsoft teams sessions per week. Participants will complete 3 sessions per week, for 4 weeks. Each session will include 6 x 6 inspirations at 80% of MIP. MIP will be measured on the supervised session day. The control group will be asked to continue as normal throughout the 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing self reported Dyspnea (Breathlessness) following COVID-19 infection over 3 months ago.
* Aged between 18 and 65

Exclusion Criteria:

* Are pregnant
* Receiving treatment following a previous cardiac event (Myocardial-infarction and Non-ST elevation MI),
* Have a dementia diagnosis,
* Have a high risk of falls,
* Have an additional chronic respiratory disease diagnosis such as (Chronic obstructive pulmonary disease) COPD or CF (cystic fibrosis)
* Are receiving respiratory muscle training
* Are receiving steroid inhaler treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in Maximal inspiratory muscle pressure (MIP) at week 4. | Baseline, and week 4
  Maximal inspiratory muscle pressure (cmH20)

SECONDARY OUTCOMES:
Change in Peak expiratory flow (PEF) at week 4. | Baseline, and week 4
  Peak expiratory flow (PEF) (l/min)
Change in Ventilatory threshold (VT) at week 4. | Baseline, and week 4
  Ventilatory threshold (VT)
Difference between Baseline Dyspnea Index score (BDI) and Transitional Dyspnea index (TDI). | Baseline, and week 4
  BDI and TDI
Change in 6 minute walk test distance at week 4 | Baseline, and week 4
  6 minute walk test difference (m)
Change in Forced ventilatory equivalent 1 second (FEV1) at week 4 | Baseline, and week 4
  Forced ventilatory equivalent 1 second (FEV1) (%)

OTHER OUTCOMES:
Change in Maximum heart rate during submaximal exercise test at week 4. | Baseline, and week 4
  Maximum heart rate during submaximal exercise (bpm)
Change in Blood pressure at week 4 | Baseline, and week 4
  Blood pressure (mmhg)
Change in Body mass index (BMI) at week 4 | Baseline, and week 4
  Body mass index (BMI) (kg/m2)
Change in Rating of perceived exertion (RPE) across submaximal exercise and 6 minute walk at week 4 | Baseline, and week 4
  Rating of perceived exertion (RPE) (Borg)
Change in Borg dyspnea scale across submaximal exercise and 6 minute walk at week 4 | Baseline, and week 4
  Borg dyspnea scale
Change in General health questionnaire (IPAQ) in week 4 | Baseline, and week 4
  General health questionnaire (IPAQ)
Change in Pittsburgh sleep quality index (PSQI) in week 4 | Baseline, and week 4
  Pittsburgh sleep quality index (PSQI)
Change in Post COVID-19 fatigue scale in week 4 | Baseline, and week 4
  Post COVID-19 fatigue scale
Change in EQ-5D-5L in week 4 | Baseline, and week 4
  EQ-5D-5L (European Quality of Life)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No